CLINICAL TRIAL: NCT05415553
Title: Inferior Oblique Muscle Belly Transposition (IOBT) Versus Inferior Oblique Muscle Recession (IO-rec) on Versions and Vertical Alignment for Primary Position Hypertropia With Inferior Oblique Overaction
Brief Title: IOBT Versus IO-Rec for Hypertropia With IOOA (IIHIOOA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Children's Hospital of Fudan University (Other); Shandong Provincial Hospital (Other Government); Shanxi Eye Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tianjin Eye Hospital (Other); Renmin Hospital of Wuhan University (Other); Xiamen Eye Center of Xiamen University (Unknown); Kunming Aier Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-IOBT
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-06

CONDITIONS: Hypertropia; Inferior Oblique Overaction
Keywords: Inferior oblique muscle belly transposition; Inferior oblique muscle recession; Inferior oblique overaction
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOBT group (Experimental): For IOBT, the whole belly of inferior oblique muscle is anchored to the sclera 5 mm behind the temporal insertion of the inferior rectus muscle.
  Interventions: Procedure: IOBT
- IO-Rec group (Active Comparator): For IO-Rec, the insertion of inferior oblique muscle is excised and anchored to the sclera 4 mm behind and 2 mm beside the temporal insertion of the inferior rectus muscle.
  Interventions: Procedure: IO-Rec

INTERVENTIONS:
Procedure: IOBT — Surgery of inferior oblique muscle belly transposition for treatment of primary position hypertropia with inferior oblique overaction
  Arms: IOBT group
Procedure: IO-Rec — Surgery of inferior oblique muscle recession for treatment of primary position hypertropia with inferior oblique overaction
  Arms: IO-Rec group

SUMMARY:
This is a multi-center, randomized double-blind controlled trial to compare the effectiveness of IOBT with IO-Rec for the treatment of hypertropia with IOOA.

Specific Aim 1 (Primary): To study the suboptimal surgical rates between IOBT and IO-Rec for the treatment of hypertropia with IOOA.

Specific Aim 2 (Secondary): To compare the surgical successful rate of IOBT with IO-Rec for the treatment of hypertropia with IOOA.

DETAILED DESCRIPTION:
Using conventional surgical procedures, such as myectomy or recession of inferior oblique muscle, higher postoperative vertical overcorrection due to contralateral concealed IOOA were observed in mild primary position hypertropia with unilateral IOOA.

To achieve better outcome, IOBT was introduced. Yang et al. firstly reported that IOBT might be a useful alternative surgical treatment for patients with primary position hypertropia of less than 5△ that was associated with IOOA. Recently, our study has reported that IOBT achieved satisfactory outcomes in patients with mild primary position vertical deviation (≤10△) with unilateral IOOA, without any risk of overcorrection of vertical deviation and contralateral IOOA. Although our results are promising, there is no enough evidence to recommend IOBT for primary position hypertropia with inferior oblique overaction. A large randomized trial is needed to compare the surgical successful rate and suboptimal surgical outcomes of IOBT with IO-Rec for primary position hypertropia with inferior oblique overaction.

The proposed trial will be conducted in 9 different study sites working in the field of pediatric ophthalmology and strabismus. Each site will have one certified surgeon to do all surgeries. For IOBT, the whole belly of inferior oblique muscle is secured with a 6-0 absorbable suture, and then anchors to the sclera 5 mm behind the temporal insertion of the inferior rectus muscle. For IO-Rec, the insertion of inferior oblique muscle is excised and secured with a 6-0 absorbable suture, and then anchors to the sclera 4 mm behind and 2 mm beside the temporal insertion of the inferior rectus muscle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4 years at the time of surgery;
* Vertical deviation (VD) in primary position (5△ ≤ VD ≤ 10△)
* IOOA for three following situations:

  1. IOOA +1 for the operative eye and IOOA - for the follow eye;
  2. IOOA +2 for the operative eye and IOOA ± for the follow eye;
  3. IOOA +2 for the operative eye and IOOA +1 for the follow eye;
* Without amblyopia

Exclusion Criteria:

* Histories of strabismus surgery or botulinum toxin injection;
* Histories of intraocular surgery or refractive surgery;
* Restrictive or paralytic strabismus;
* Ocular disease other than strabismus or refractive error;
* Craniofacial malformations affecting the orbits;
* Significant neurological disorders

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Suboptimal surgical rate | at 12 months
  Suboptimal surgical cases/total cases. Suboptimal surgical outcomes include vertical undercorrection, vertical overcorrection and antielevation syndrome.

SECONDARY OUTCOMES:
Surgical successful rate | at 12 month
  Surgical successful cases/total cases. The successful criterion is without any vertical deviation in primary position at distance and without IOOA postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.

REFERENCES:
- [Background] Bahl RS, Marcotty A, Rychwalski PJ, Traboulsi EI. Comparison of inferior oblique myectomy to recession for the treatment of superior oblique palsy. Br J Ophthalmol. 2013 Feb;97(2):184-8. doi: 10.1136/bjophthalmol-2012-301485. Epub 2012 Nov 30. PMID 23203704
- [Background] Alajbegovic-Halimic J, Zvizdic D, Sahbegovic-Holcner A, Kulanic-Kuduzovic A. Recession Vs Myotomy-Comparative Analysis of Two Surgical Procedures of Weakening Inferior Oblique Muscle Overaction. Med Arch. 2015 Jun;69(3):165-8. doi: 10.5455/medarh.2015.69.165-168. Epub 2015 Jun 10. PMID 26261384
- [Background] Nabie R, Raoufi S, Hassanpour E, Nikniaz L, Kharrazi B, Mamaghani S. Comparing graded anterior transposition with myectomy in primary inferior oblique overaction - A clinical trial. J Curr Ophthalmol. 2019 May 8;31(4):422-425. doi: 10.1016/j.joco.2019.04.002. eCollection 2019 Dec. PMID 31844794
- [Background] Akbari MR, Sadrkhanlou S, Mirmohammadsadeghi A. Surgical Outcome of Single Inferior Oblique Myectomy in Small and Large Hypertropia of Unilateral Superior Oblique Palsy. J Pediatr Ophthalmol Strabismus. 2019 Jan 23;56(1):23-27. doi: 10.3928/01913913-20180925-03. Epub 2018 Oct 26. PMID 30371917
- [Background] Hendler K, Pineles SL, Demer JL, Rosenbaum AL, Velez G, Velez FG. Does inferior oblique recession cause overcorrections in laterally incomitant small hypertropias due to superior oblique palsy? Br J Ophthalmol. 2013 Jan;97(1):88-91. doi: 10.1136/bjophthalmol-2012-302006. Epub 2012 Nov 10. PMID 23143910
- [Background] Bhatta S, Auger G, Ung T, Burke J. Underacting inferior oblique muscle following myectomy or recession for unilateral inferior oblique overaction. J Pediatr Ophthalmol Strabismus. 2012 Jan-Feb;49(1):43-8. doi: 10.3928/01913913-20110208-02. Epub 2011 Feb 15. PMID 21323243
- [Background] Yang S, Guo X, Tien DR. Inferior Oblique Belly Transposition for Small Angle Hypertropia With Inferior Oblique Overaction: A Pilot Study. J Pediatr Ophthalmol Strabismus. 2018 Jan 1;55(1):43-46. doi: 10.3928/01913913-20170801-04. Epub 2017 Oct 9. PMID 28991348
- [Background] Zhu W, Wang X, Jiang C, Ling L, Wu L, Zhao C. Effect of inferior oblique muscle belly transposition on versions and vertical alignment in primary position. Graefes Arch Clin Exp Ophthalmol. 2021 Nov;259(11):3461-3468. doi: 10.1007/s00417-021-05240-x. Epub 2021 Jun 18. PMID 34142185
- [Background] Tomarchio S, Sabetti L, Tomarchio M, Berarducci A. New surgical intervention for the weakening of the inferior oblique muscle: equatorial scleral anchor. J Pediatr Ophthalmol Strabismus. 2015 Jan-Feb;52(1):58-60. doi: 10.3928/01913913-20141230-09. PMID 25643372
- [Background] Kasem M, Metwally H, El-Adawy IT, Abdelhameed AG. Retro-equatorial inferior oblique myopexy for treatment of inferior oblique overaction. Graefes Arch Clin Exp Ophthalmol. 2020 Sep;258(9):1991-1997. doi: 10.1007/s00417-020-04742-4. Epub 2020 May 27. PMID 32462341
- [Background] Shipman T, Burke J. Unilateral inferior oblique muscle myectomy and recession in the treatment of inferior oblique muscle overaction: a longitudinal study. Eye (Lond). 2003 Nov;17(9):1013-8. doi: 10.1038/sj.eye.6700488. PMID 14704751